CLINICAL TRIAL: NCT06864910
Title: Brain Connectivity in Mild Cognitive Impairment and Alzheimer's Disease: A Resting and Task-based fMRI-MEG Study Examining Alterations in Functional Connectivity Following Treatment With Transcranial Current Stimulation (tDCS)
Brief Title: Brain Functional Changes Accompany Modulatory Effects of Transcranial Direct Current Stimulation in Cognitive Impairment
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health and Neuro Sciences, India (Other)
Responsible Party: Principal Investigator, John P John, Professor of Psychiatry, National Institute of Mental Health and Neuro Sciences, India
Other Study IDs: DST-CSI/002/208/2018/01156; DST/CSRI/2017/249 (G) 28.08.18 (Other Grant/Funding Number: Department of Science and Technology, Government of India)
Record Dates: First submitted 2025-02-14; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Cognitive Impairment
Keywords: transcranial Direct current Stimulation; Alzheimer Disease; Mild Cognitive Impairment; functional Magnetic Resonance Imaging; Magnetoencephalography
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- early Alzheimer's Disease (AD): The early AD group comprised of patients with Mild Cognitive Impairment (MCI) and mild Alzheimer's Disease (AD)
  Interventions: Device: anodal transcranial Direct Current Stimulation

INTERVENTIONS:
Device: anodal transcranial Direct Current Stimulation — Transcranial direct current stimulation was administered following standard procedures using a neuroConn DC-Stimulator Plus device (neuroCare Group GmbH, Munich, Germany) with the anode placed at F3 (left DLPFC) and the cathode over the right supraorbital region (Fp2) using 5x7cm electrodes. The anodal tDCS intervention involved daily sessions (between 10-11 a.m.) for 10 consecutive days, wherein a direct current (DC) of 2 mA was administered for 20 minutes (with additional ramp-up and ramp-down phase of 20 seconds each at the beginning and end of the session respectively), adhering to stringent safety measures . None of the participants reported significant adverse effects.

SUMMARY:
The goal of this observational study was to examine the brain functional alterations accompanying cognitive modulatory effect of anodal transcranial Direct Current Stimulation (tDCS) in sample patients with early Alzheimer's Disease (AD), registered under Geriatric Clinic and Services at NIMHANS, and who were initiated on tDCS for cognitive enhancement. Further, to explore the potential beneficial effect of tDCS, the investigators offered the intervention to the first 40 consenting patients from the amnestic Mild Cognitive Impairment (aMCI) (n=21) and mild AD (n=19) samples. The changes in functional connectivity/activations associated with diminished cognitive functions were examined using functional magnetic resonance imaging (fMRI) and magnetoencephalography (MEG), between pre- and post-tDCS intervention. The administration of tDCS followed the standard procedures using a neuroConn DC-Stimulator Plus device (neuroCare Group GmbH, Munich, Germany) with the anode placed at F3 (left DLPFC) and the cathode over the right supraorbital region (Fp2) using 5x7cm electrodes. The anodal tDCS intervention involved daily sessions (between 10-11 a.m.) for 10 consecutive days, wherein a direct current (DC) of 2 mA was administered for 20 minutes (with additional ramp-up and ramp-down phase of 20 seconds each at the beginning and end of the session respectively), adhering to stringent safety measures.

DETAILED DESCRIPTION:
As apriori registration was not done before the initiation of the study and all the participants already underwent tDCS intervention, the investigators are herewith submitting the protocol of the study retrospectively following the completion of the project. This study was conducted at the National Institute of Mental Health and Neurosciences (NIMHANS), Bengaluru, India, with the approval of the NIMHANS Institutional Ethics Committee.

Study Sample: All consenting participants of both sexes (age range: 55 - 84 years) meeting the inclusion and exclusion criteria (see below), who consecutively attended the outpatient services of the Geriatric Clinic and Services (GCS), NIMHANS from August 2019 to December 2022 with memory complaints were recruited in this study with their signed informed consent. Only right-handed individuals were recruited as assessed using the Edinburgh Handedness Inventory (EHI). Participants were screened to ensure that only those with optimal hearing and visual acuity were recruited. The clinical diagnoses of MCI and mild AD made by clinicians at the GCS at NIMHANS were confirmed using the National Institute on Ageing - Alzheimer's Association (NIA-AA) diagnostic criteria and Clinical Dementia Rating [CDR] (CDR scores of 0.5 for MCI and 1 for mild AD). Participants with CDR scores above 1 were excluded from this study. Other exclusion criteria included concurrent medical conditions like hypothyroidism, hypercalcemia, vitamin B12 deficiency, uncontrolled hypertension and diabetes, neurosyphilis, normal pressure hydrocephalus, subdural hematoma, etc., requiring initiation of medical/surgical interventions and/or titration of medications; pre-existing major psychiatric and neurological illnesses, such as schizophrenia spectrum disorders, bipolar affective disorder, major depressive disorder, obsessive-compulsive disorder, substance dependence, intellectual disability disorder, Parkinson's disease and related disorders, stroke, epilepsy, and other chronic neurological/neurodegenerative disorders, and significant head injury; and current usage of antipsychotics, antidepressants, and benzodiazepines. Forty patients (19 MCI and 21 mild AD) consented to participate in the study and completed the tDCS intervention protocol, which comprised daily 20-minute tDCS sessions for 10 days. All participants underwent detailed neuropsychological assessments, resting-state functional magnetic resonance imaging (rsfMRI), task-based functional magnetic resonance imaging (tbfMRI) as well as resting state magnetoencephalography (rsMEG) following tDCS intervention.

Neuropsychological Battery for Elderly (NNB-E): This battery includes tests of episodic memory, executive functions, attention, visuospatial function, and parietal focal signs and required 1.5 hours to administer and score. Assessments were carried out at baseline (pre-tDCS) and after completion of the last tDCS session (post-tDCS). These pre- and post-tDCS assessments were conducted in a way that prevented the same researcher from doing both tests for a particular participant. Additionally, the person conducting the post-tDCS assessment was blind to the results of the pre-assessment. Two different forms were used for the pre-and post-tDCS assessments of a participant to avoid practice effects. Shapiro Wilk test was performed to check the normality distribution of the differences between pre- and post-tDCS scores for each sub-test (n=26) of NNB-E. Accordingly, paired t-tests and Wilcoxon signed rank tests were carried out respectively for normally and non-normally distributed sub-test scores to look for significant effects of tDCS intervention.

Magnetic Resonance Imaging (MRI): The MRIs were acquired on a 3Tesla Philips Ingenia CX (Philips Healthcare, Netherlands) scanner with a 32-channel phased-array head coil. During rs-fMRI acquisition, the participants were instructed to remain physically and mentally relaxed with their eyes open and not focus on anything particular. These functional MR images corresponding to each participant were visually examined for scanner or acquisition-related artifacts. The rs-fMRI data of one participant each from the MCI and mild AD groups showed more than 5% intensity variation in two consecutive volumes indicating poor quality of functional images due to motion artifacts validated using Derivative of root mean square VARiance over voxelS (DVARS). After the exclusion of both pre- and post-rsfMRI scans of these two participants, the data of the remaining 38 participants (n=18 in the MCI group and n=20 in the mild AD group) were further analyzed. The seed for the seed-to-voxel resting state functional connectivity (S2V-rsFC) analysis was set using the Harvard cortical atlas, as the left middle frontal gyrus (lMFG), corresponding to the left DLPFC, the site of the anodal tDCS. The analysis between pre- and post-tDCS intervention was performed using the spherical mask of lMFG as 'seed' and the whole-brain volume for 'voxels'. Two-tailed parametric statistics were implemented to obtain the results using a cluster-level extent threshold (p-FDR corrected) with voxel threshold at p < 0.001 (p-uncorrected) and cluster threshold at p < 0.05 (p-corrected).

A novel episodic memory paradigm, comprising two tasks: an incidental encoding task and an intentional retrieval task, was used for tb-fMRI acquisition. In the incidental encoding task, the participants were instructed on each trial to indicate using a button press whether the presented visual images were of living or non-living objects. In the intentional retrieval task, the instruction for each trial was to indicate using a button press, whether the presented visual images were seen before (memory images, MI) or not seen before (non-memory images, nMI). The optimal number of trials for the incidental encoding task (living objects: 55; non-living objects: 55; fixation cross: 56) and the intentional retrieval task (memory images, MI: 55; non-memory images, nMI: 55; fixation cross: 56) was estimated using the fMRI stimulator to maximize the predictable variance between the three trial classes for each of the two tasks. Only the participants showing more than 60% performance accuracy on both incidental encoding and intentional retrieval were analyzed. Task-based fMRI data pre-processing and analyses of remaining participants with early AD (n=30; MCI=15, mild AD=15) were carried out using FMRI Expert Analysis Tool (FEAT) Version 6.00 of FMRIB Software Library (FSL), implementing high-quality model-based fMRI data analysis. Z (Gaussianised T/F) statistical images were thresholded non-parametrically using clusters determined by Z > 2.3 and a corrected cluster significance threshold of P=0.05.

Magnetoencephalography (MEG): The pre- and post- rsMEG data were acquired using the Elekta Neuromag® TRIUX™ MEG Scanner. Two participants (1 in the MCI sample and 1 in the mild AD sample) opted out of taking part in MEG acquisition, and four participants (3 in the MCI sample and 1 in the mild AD sample) did not participate in post-MEG scans; MEG data of the remaining participants with early AD (n=34; MCI=15, mild AD=19) were further preprocessed. The resting eyes closed MEG recordings were carried out in a sitting position employing the following protocol: sampling rate 2000 Hz, empty room recording=2 minutes, resting-state MEG=15 minutes. EEG data were acquired concurrently to ensure that the participants were alert and relaxed during the recording. Electrocardiogram (ECG), electromyography (EMG), and electrooculogram (EOG) were acquired to remove the heart, muscle, and ocular artifacts, respectively. Quality control (QC) of the MEG data was done using MaxfilterTM (ver 2.2), a built-in software for the ELEKTA/Neuromag system. Suppression of interference due to environmental and periodic artifacts was carried out using the spatiotemporal signal space separation (tSSS) method. Using the Welch method, a power spectrum analysis was performed on 5 minutes of artifact-free MEG recording. Extracted power spectrum density (PSD) values for neural oscillations covered canonical frequency bands [delta (2-4 Hz), theta (4-8 Hz), alpha (8-12 Hz), beta (13-30 Hz), gamma (30-60 Hz) and gamma2 (60-90 Hz)]. A paired T-test was performed between the pre- and post-tDCS values of normalized PSD, correcting for multiple [permutation testing (1000 randomizations), Monte Carlo method] comparisons (FDR-corrected), controlling for time and frequency.

The dependence between the phase of low-frequency oscillations (fP) and the amplitude of high-frequency rhythms (fA) was quantified using phase amplitude coupling (PAC). The coupling strength for each participant was estimated using time-resolved PAC (tPAC), which shows the least relative error. The tPAC was estimated by searching for the fP oscillation with the strongest PAC to fA bursts, over a time window, which slides on the input MEG data. A 10-second epoch length was used for analysis, and since the fP band of interest was between 4-8 Hz, three full cycles of the fP band were chosen to produce a sliding window length of 0.75 seconds. The average comodulograms were extracted using tPAC maps of all the patients with MCI (n=15) and mild AD (n=19) in the left entorhinal cortex which plays a critical role in episodic memory and is vulnerable to early pathophysiology in AD. A paired t-test was performed outside this software using MATLAB® (https://www.mathworks.com) to find out the significant (FDR-corrected p < 0.05) difference in coupling strength between phase of low frequencies (4-8 Hz) and amplitude of high frequencies (30-90 Hz) correcting for multiple comparisons across time and frequency.

ELIGIBILITY:
Patients with Mild Cognitive Impairment and mild Alzheimer's Disease

Inclusion Criteria:

* Elderly aged 55 years or above
* Both genders
* Only right handed individuals
* Elderly with a diagnosis of Minimal Cognitive Impairment and Mild AD according to National institute of Ageing -Alzheimer's Association (NIAAA) diagnostic Criteria and 0.5 for MCI and 1 according to CDR criteria.
* Informed consent

Exclusion Criteria:

* Elderly with more advanced dementia (CDR >1)
* Patients on medications like antipsychotics, antidepressants and benzodiazepines (some of patients).
* Patient with comorbid clinical conditions like hypothyroidism, hypercalcemia, vitamin B12 deficiency, niacin deficiency, neurosyphilis, normal pressure hydrocephalus or subdural haematoma.
* Persons with other mental disorders like schizophrenia and related disorder, bipolar affective disorder, severe depression, obsessive compulsive disorder, substance dependence and mental retardation.
* History of neurological illness like stroke, epilepsy, head injury with significant loss of consciousness or other chronic neurological/ neurodegenerative conditions.

Elderly Cognitively Healthy Comparison group (n=50)

Inclusion criteria

* Elderly aged 55 years or above (age, gender and education matched with Dementia subjects)
* Persons without MCI/AD (NIAAA Criteria)
* Both genders, only right handed individuals.
* Informed consent Exclusion criteria
* Elderly with MCI or dementia (CDR ≥0.5)
* Patients on medications like antipsychotics, antidepressants and benzodiazepines (some of patients).
* Patient with comorbid clinical conditions like hypothyroidism, hypercalcemia, vitamin B12 deficiency, niacin deficiency, neurosyphilis, normal pressure hydrocephalus or subdural haematoma.
* Persons with other mental disorders like schizophrenia and related disorder, bipolar affective disorder, severe depression, obsessive compulsive disorder, substance dependence and mental retardation.

History of neurological illness like stroke, epilepsy, head injury with significant loss of consciousness or other chronic neurological/ neurodegenerative conditions.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males and Females
Study Population: All consecutive patients aged 55 and above attending the Geriatric Clinic and Services at NIMHANS with memory complaints who fulfil the following inclusion and exclusion criteria will be considered for recruitment into the study. Those diagnosed as Minimal Cognitive Impairment or Mild Alzheimer's Dementia by two consultants according to National Institute of Aging and Alzheimer's Association criteria and a Clinical Dementia Rating (CDR) of 0.5 for MCI and 1 for Mild AD would be recruited. Consenting cognitively healthy elderly subjects matched for age and gender to the above with CDR < 0.5 would be parallely recruited.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Magnetic Resonance Imaging | After the completion of 10 sessions of tDCS (one session per day) spanning across a maximum of 14 days
  The resting state functional connectivity, incidental encoding and intentional retrieval task based activation were the primary outcome measures of MRI.
Magnetoencephalography | After the completion of 10 sessions of tDCS (one session per day) spanning across a maximum of 14 days
  The power of alpha, beta, theta and gamma bandwidths, phase of theta waves and amplitude of gamma band coupling in the left entorhinal cortex were calculated as primary outcome measure of magnetoencephalography
Cognitive assessments | After the completion of 10 sessions of tDCS (one session per day) spanning across a maximum of 14 days
  The output of NIMHANS Neuropsychological Battery for Elderly (NNB-E) measuring tests of episodic memory, executive functions, attention, visuospatial function, and parietal focal signs were noted as primary outcome measures of the cognitive assessments used in this study.

CONTACTS AND LOCATIONS:
Overall Officials: John P John, M.D., Principal Investigator — National Institute of Mental Health and Neuro Sciences, India
Locations (2):
- India (2):
  - National Institute of Mental Health and Neurosciences (NIMHANS), Bengaluru, Karnataka
  - National Institute of Mental Health and Neurosciences, Bengaluru, Karnataka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodriguez GA, Barrett GM, Duff KE, Hussaini SA. Chemogenetic attenuation of neuronal activity in the entorhinal cortex reduces Abeta and tau pathology in the hippocampus. PLoS Biol. 2020 Aug 21;18(8):e3000851. doi: 10.1371/journal.pbio.3000851. eCollection 2020 Aug. PMID 32822389
- [Background] Jacobs J, Kahana MJ, Ekstrom AD, Fried I. Brain oscillations control timing of single-neuron activity in humans. J Neurosci. 2007 Apr 4;27(14):3839-44. doi: 10.1523/JNEUROSCI.4636-06.2007. PMID 17409248
- [Background] Tadel F, Baillet S, Mosher JC, Pantazis D, Leahy RM. Brainstorm: a user-friendly application for MEG/EEG analysis. Comput Intell Neurosci. 2011;2011:879716. doi: 10.1155/2011/879716. Epub 2011 Apr 13. PMID 21584256
- [Background] Uusitalo MA, Ilmoniemi RJ. Signal-space projection method for separating MEG or EEG into components. Med Biol Eng Comput. 1997 Mar;35(2):135-40. doi: 10.1007/BF02534144. No abstract available. PMID 9136207
- [Background] Behzadi Y, Restom K, Liau J, Liu TT. A component based noise correction method (CompCor) for BOLD and perfusion based fMRI. Neuroimage. 2007 Aug 1;37(1):90-101. doi: 10.1016/j.neuroimage.2007.04.042. Epub 2007 May 3. PMID 17560126
- [Background] Friston KJ, Williams S, Howard R, Frackowiak RS, Turner R. Movement-related effects in fMRI time-series. Magn Reson Med. 1996 Mar;35(3):346-55. doi: 10.1002/mrm.1910350312. PMID 8699946
- [Background] Andersson JL, Skare S, Ashburner J. How to correct susceptibility distortions in spin-echo echo-planar images: application to diffusion tensor imaging. Neuroimage. 2003 Oct;20(2):870-88. doi: 10.1016/S1053-8119(03)00336-7. PMID 14568458
- [Background] Whitfield-Gabrieli S, Nieto-Castanon A. Conn: a functional connectivity toolbox for correlated and anticorrelated brain networks. Brain Connect. 2012;2(3):125-41. doi: 10.1089/brain.2012.0073. Epub 2012 Jul 19. PMID 22642651
- [Background] Power JD, Barnes KA, Snyder AZ, Schlaggar BL, Petersen SE. Spurious but systematic correlations in functional connectivity MRI networks arise from subject motion. Neuroimage. 2012 Feb 1;59(3):2142-54. doi: 10.1016/j.neuroimage.2011.10.018. Epub 2011 Oct 14. PMID 22019881
- [Background] Smith SM, Jenkinson M, Woolrich MW, Beckmann CF, Behrens TE, Johansen-Berg H, Bannister PR, De Luca M, Drobnjak I, Flitney DE, Niazy RK, Saunders J, Vickers J, Zhang Y, De Stefano N, Brady JM, Matthews PM. Advances in functional and structural MR image analysis and implementation as FSL. Neuroimage. 2004;23 Suppl 1:S208-19. doi: 10.1016/j.neuroimage.2004.07.051. PMID 15501092
- [Background] Taulu S, Simola J. Spatiotemporal signal space separation method for rejecting nearby interference in MEG measurements. Phys Med Biol. 2006 Apr 7;51(7):1759-68. doi: 10.1088/0031-9155/51/7/008. Epub 2006 Mar 16. PMID 16552102
- [Background] Snodgrass JG, Vanderwart M. A standardized set of 260 pictures: norms for name agreement, image agreement, familiarity, and visual complexity. J Exp Psychol Hum Learn. 1980 Mar;6(2):174-215. doi: 10.1037//0278-7393.6.2.174. PMID 7373248
- [Background] Sternberg S. High-speed scanning in human memory. Science. 1966 Aug 5;153(3736):652-4. doi: 10.1126/science.153.3736.652. PMID 5939936
- [Background] Gardiner JM. Functional aspects of recollective experience. Mem Cognit. 1988 Jul;16(4):309-13. doi: 10.3758/bf03197041. No abstract available. PMID 3210971
- [Background] Parekh P, Bhalerao GV, Rao R, Sreeraj VS, Holla B, Saini J, Venkatasubramanian G, John JP, Jain S; ADBS Consortium. Protocol for magnetic resonance imaging acquisition, quality assurance, and quality check for the Accelerator program for Discovery in Brain disorders using Stem cells. Int J Methods Psychiatr Res. 2021 Sep;30(3):e1871. doi: 10.1002/mpr.1871. Epub 2021 May 7. PMID 33960571
- [Background] Brunoni AR, Amadera J, Berbel B, Volz MS, Rizzerio BG, Fregni F. A systematic review on reporting and assessment of adverse effects associated with transcranial direct current stimulation. Int J Neuropsychopharmacol. 2011 Sep;14(8):1133-45. doi: 10.1017/S1461145710001690. Epub 2011 Feb 15. PMID 21320389
- [Background] Tripathi R, Kumar JK, Bharath S, Marimuthu P, Varghese M. Clinical validity of NIMHANS neuropsychological battery for elderly: A preliminary report. Indian J Psychiatry. 2013 Jul;55(3):279-82. doi: 10.4103/0019-5545.117149. PMID 24082250
- [Background] McKhann GM, Knopman DS, Chertkow H, Hyman BT, Jack CR Jr, Kawas CH, Klunk WE, Koroshetz WJ, Manly JJ, Mayeux R, Mohs RC, Morris JC, Rossor MN, Scheltens P, Carrillo MC, Thies B, Weintraub S, Phelps CH. The diagnosis of dementia due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):263-9. doi: 10.1016/j.jalz.2011.03.005. Epub 2011 Apr 21. PMID 21514250
- [Background] Albert MS, DeKosky ST, Dickson D, Dubois B, Feldman HH, Fox NC, Gamst A, Holtzman DM, Jagust WJ, Petersen RC, Snyder PJ, Carrillo MC, Thies B, Phelps CH. The diagnosis of mild cognitive impairment due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):270-9. doi: 10.1016/j.jalz.2011.03.008. Epub 2011 Apr 21. PMID 21514249

DOCUMENTS (1):
  • Informed Consent Form (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT06864910/ICF_000.pdf